CLINICAL TRIAL: NCT04240782
Title: Market to MyPlate: A Cluster Randomized Trial Investigating the Impact of a Nutrition and Hands-On Cooking Intervention on Dietary, Cooking, and Shopping Behaviors
Brief Title: Market to MyPlate: Investigating the Impact of a Nutrition and Hands-On Cooking Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17806
Record Dates: First submitted 2019-12-19; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-12

CONDITIONS: Fruit and Vegetable Consumption; Cooking Frequency
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education with Produce Allocations (Experimental): Participants will attend nutrition education and hands-on cooking classes with weekly produce allocations from a local farm.
  Interventions: Behavioral: Nutrition and hands on cooking classes for parents and their children; Behavioral: Produce allocations
- Education only (Experimental): Participants will attend nutrition education and hands-on cooking classes (with produce coupons provided after intervention).
  Interventions: Behavioral: Nutrition and hands on cooking classes for parents and their children
- Control group (No Intervention): Participants will receive a delayed intervention once the study period is over.

INTERVENTIONS:
Behavioral: Nutrition and hands on cooking classes for parents and their children — The adults and children will learn how to prepare the fresh produce during an age appropriate, evidence-based, family cooking school. The class will provide participants with a no-cost, low-risk incentive to try new vegetables, and will empower them to build healthier lives through nutrient-rich, locally sourced meals. Participants will also receive nutrition education and information on how they can integrate local produce into their food budget. One of the class sessions will focus solely on how to budget for healthy food, comparison shop, and make the most of their food dollars. Participants will learn how to use their SNAP benefits at local farmers markets.
  Arms: Education only; Education with Produce Allocations
Behavioral: Produce allocations — Participants will also receive a produce allocation from a local farm during each session of the class.
  Arms: Education with Produce Allocations

SUMMARY:
Recent peer-reviewed research indicates that low-income families are at higher risk for unhealthy dietary intake and associated poor health outcomes. Interventions that teach individuals from low-income families about cooking and healthy eating are warranted to improve overall dietary behaviors. The purpose of this study is to evaluate the impact of the Market to MyPlate Program on participants' reported cooking, shopping, and dietary behaviors using a cluster randomized trial design, where class cohorts are randomly assigned to education with produce allocations, education only, or control conditions. A secondary aim is to collect program feedback and better understand facilitators and barriers to farmer's market use and food waste reduction.

ELIGIBILITY:
Inclusion Criteria:

* Recruited from SNAP-Ed eligible site (site where the majority of participants are eligible for US food assistance programs)
* Must be 18 years or older, or parent of any age with child(ren) to participate in data collection (all ages including children could participate in intervention)

Exclusion Criteria:

• Participated in an Extension nutrition education program in the last year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Self-reported vegetable consumption | 7 weeks
  Survey asks participants to self-report how frequently they consume fruits and vegetables.
self-reported shopping behaviors | 7 weeks
  Survey asks participants to self-report how frequently they compare food prices, make shopping lists, and plan meals before grocery shopping.
self-reported cooking behaviors | 7 weeks
  Survey asks participants to self-report how frequently they cook dinner at home.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided